CLINICAL TRIAL: NCT01041976
Title: Supported Employment: Motivational Enhancement for Entry and Outcome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7306-R
Record Dates: First submitted 2009-12-31; First posted 2010-01-05 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Psychotic Disorders; Bipolar Disorder; Unemployment
Keywords: Veterans; Vocational Rehabilitation
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder | interventions — Palliative Care; Educational Status; Salvage Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adapted Motivational Interviewing (AMI) (Experimental): Veterans assigned to the AMI condition will be scheduled for up to 6 sessions over 6 months. Up to 3 of these 6 sessions will be joint sessions with the Veteran's significant other (if available). Sessions will utilize a variety of motivational enhancement strategies including evocative questions, importance and confidence scales, collaborative problem solving, and planning.
  Interventions: Behavioral: Adapted Motivational Interviewing (AMI)
- Support and Education for Recovery (SER) (Placebo Comparator): Veterans assigned to the control condition will be seen for 6 sessions over 6 months of basic support and education about VA and non-VA psychiatric rehabilitation and recovery services. Up to 3 of these 6 sessions will be joint sessions with the Veteran's significant other (if available). The session topics include information about Bedford VA and Boston VA recovery services, as well as those offered by local non-profits.
  Interventions: Behavioral: Support and Education for Recovery (SER)

INTERVENTIONS:
Behavioral: Adapted Motivational Interviewing (AMI) — Veterans assigned to the AMI condition will be scheduled for up to 6 sessions over 6 months. Up to 3 of these 6 sessions will be joint sessions with the Veteran's significant other (if available). Sessions will utilize a variety of motivational enhancement strategies including evocative questions, importance and confidence scales, collaborative problem solving, and planning.
  Arms: Adapted Motivational Interviewing (AMI)
Behavioral: Support and Education for Recovery (SER) — Veterans assigned to the control condition will be seen for 6 sessions over 6 months of basic support and education about VA and non-VA psychiatric rehabilitation and recovery services. Up to 3 of these 6 sessions will be joint sessions with the Veteran's significant other (if available). The session topics include information about Bedford VA and Boston VA recovery services, as well as those offered by local non-profits.
  Arms: Support and Education for Recovery (SER)

SUMMARY:
The purpose of this study is to compare 6 monthly counseling sessions to 6 monthly information sessions on Veterans' decisions to (a) participate in vocational rehabilitation services and (b) become employed.

DETAILED DESCRIPTION:
Approximately 85-90% of those with serious mental illness are unemployed (9, 10). This level of unemployment exists despite the finding that, among people who have a psychiatric disability and are unemployed, 55-61% desire employment, with the total reaching 75% when concern about losing benefits was taken into account (1, 2). The rewards of employment for adults with SMI are greater than simply an increase in financial resources. Studies have found that people with serious mental illness who worked competitively scored higher on measures of self-esteem, satisfaction with finances, leisure, and overall life satisfaction compared to those worked little or not at all (11). Supported employment (SE) has been more effective than any other vocational rehabilitation approach for this population (3, 4) and the VA has mandated that SE be integrated into all current VHA Compensated Work Therapy (CWT) programs (VHA Directive 2007-005). Two areas of concern include (a) national utilization of SE services is low (13), and (b) the percentage of SE participants who obtain at least one job during the studies averages 56% even though everyone who enters the program expressed an interest in working (13).

Motivational interviewing (MI) is an evidence-based practice that has been effective in enhancing a range of clinical services (6), but has just recently been applied to employment and vocational services by Drebing et al. (7) and Glynn et al (8).

The proposed project is a randomized trial of Adapted Motivational Interviewing for Supported Employment (AMI-SE) provided to Veterans and their significant others (family members or key friends) in order to address the internal and external barriers to the Veteran enrolling in supported employment and returning to work.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to receive VA services
* Diagnosis of serious mental illness: schizophrenia, schizoaffective, psychosis NOS, bipolar disorder, or depression with psychotic features
* Currently unemployed
* Not currently enrolled in Supported Employment services
* Expects to stay within 100 miles of Bedford, MA for the next 18 months
* Has a significant other (friend or family member) who is also willing to participate (a criterion required only from March 2011 to March 2012 of the recruitment period)

Exclusion Criteria:

* Currently in prison
* Not able to provide informed consent
* Not able to speak and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-01; Primary Completion 2014-05 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Mueller, PhD MSEd, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a variety of clinics at the Edith Nourse Rogers Memorial VA Hospital including: the Psychosocial Rehabilitation and Recovery Center, Mental Health Intensive Case Management (MHICM), outpatient Prolixin and Clozaril clinics, VA Supported Housing (VASH), and the psychiatric inpatient unit.
Pre-assignment Details: 168 participants enrolled, 115 veterans+53 family/key friends willing to participate, a criterion only for 3/2011-3/2012 recruitment. Veterans completed screening interview and if eligible completed the informed consent process and baseline interview. During 1st session with individual research clinician 84 Veterans were randomized to AMI or SER.
Period: Overall Study
Arm/Group | Adapted Motivational Interviewing (AMI) | Support and Education for Recovery (SER)
Started | 42 | 42
6 Month Follow-up | 39 | 41
12 Month Follow-up | 37 | 38
18 Month Follow-up | 37 | 38
Completed | 37 | 38
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Incarceration | 2 | 0
Not completed — Death | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapted Motivational Interviewing (AMI) | Support and Education for Recovery (SER) | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (11.0) | 53.0 (8.6) | 53.0 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 38 | 42 | 80
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian/Alaskan | 0 | 1 | 1
  Asian/Pacific Islander | 1 | 0 | 1
  Black/African-American | 9 | 6 | 15
  White | 27 | 28 | 55
  Multi-racial | 2 | 5 | 7
  Hispanic/Latino, White | 3 | 2 | 5
  Hispanic/Latino, Black | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Participation in Vocational Rehabilitation Services
Description: Yes/No: Did veteran complete an intake for a VA Supported Employment program at any time from randomization to 18 month follow-up.
  Outcome: Number of participants who completed an intake for VA Supported Employment program at any time from randomization to 18 month follow-up.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Adapted Motivational Interviewing (AMI) | Support and Education for Recovery (SER)
Number analyzed (Participants) | 42 | 42
participants | 19 | 3
Statistical Analysis 1: Comparison: Adapted Motivational Interviewing (AMI) vs Support and Education for Recovery (SER); Test type: Superiority or Other; p < 0.001, Chi-squared

2. Secondary Outcome: Employment
Description: Yes/No: Did veteran work at least one day in a competitive job at any time from randomization to 18 month follow-up.
  Outcome: Number of participants who worked at least one day in a competitive job at any time from randomization to 18 month follow-up.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Adapted Motivational Interviewing (AMI) | Support and Education for Recovery (SER)
Number analyzed (Participants) | 42 | 42
participants | 12 | 4
Statistical Analysis 1: Comparison: Adapted Motivational Interviewing (AMI) vs Support and Education for Recovery (SER); Test type: Superiority or Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the time period beginning with informed consent and ending with the 18 month follow-up for each participant.
Arm/Group | Adapted Motivational Interviewing (AMI) | Support and Education for Recovery (SER)
Serious Adverse Events (participants affected / at risk) | 15/42 | 20/42
Other Adverse Events (participants affected / at risk) | 0/42 | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapted Motivational Interviewing (AMI) (N=42) | Support and Education for Recovery (SER) (N=42)
Psychiatric Hospitalization (Psychiatric disorders) | 13 (22) | 14 (38)
Medical Hospitalization (General disorders) | 5 (7) | 9 (13)
Death (General disorders) | 0 (0) | 4 (4)
Arrest & Incarceration (Social circumstances) | 2 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapted Motivational Interviewing (AMI) (N=42) | Support and Education for Recovery (SER) (N=42)
Emergency Room Visit (General disorders) | 0 (0) | 2 (3)
Transfer Within Hospital (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes